CLINICAL TRIAL: NCT03301402
Title: A Randomized Controlled Trial of Air Purifier to Improve Endothelial Function and Carotid Intima Thickness in Older Diabetic People With Cognitive Impairment
Brief Title: Air Purifier to Improve Endothelial Function and Carotid Intima Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017.304
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Endothelial Function; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filter (Active Comparator)
  Interventions: Device: Air purifier
- No filter (No Intervention)

INTERVENTIONS:
Device: Air purifier — Air purifier with filter at automatic mode on all time
  Arms: Filter

SUMMARY:
Background: There is epidemiological evidence or link ambient air pollution exposure to the incidence of dementia.

Aims or hypotheses: It is hypothesized that reduction in indoor pollutants from air purification improves endothelial function and carotid intima thickness in older diabetic people with cognitive impairment.

Subjects and method: People with clinically diagnosis mild cognitive impairment or early dementia will be recruited. After obtaining written consent, the subjects will be assessed cognitive function and arterial health. After baseline measurements, the subjects are randomly assigned to have either filter or no filter installed in the air purifier. The air purifier will be placed in living room of the household of the subject for one year. At one year, the measurements will be repeated.

Statistical analysis: Intention to treat analysis will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic people
* Mild cognitive impairment or early dementia

Exclusion Criteria:

* Current smoker
* The presence of a smoker in the household
* The absence of a reliable family caregiver
* The lack of mental capacity to give informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
FMD% | 12 months
  Endothelial function will be assessed by Flow mediated dilatation of brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong